CLINICAL TRIAL: NCT05934682
Title: Latin American Surgical Outcomes Study in Pediatric Patients
Acronym: LASOS-Peds
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria José Carvalho Carmona, Associate Professor, University of Sao Paulo
Other Study IDs: LASOS-Peds
Record Dates: First submitted 2023-06-19; First posted 2023-07-07 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Complications; Children; Neonate; Infant; Anesthesia
MeSH Terms: conditions — Postoperative Complications | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children submitted to surgery: We will follow children submitted to surgery until hospital discharge or until 30 days after surgery.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — All children submitted to surgery will be followed until hospital discharge or 30 days postoperatively.

SUMMARY:
This prospective, international, multicenter observational study will include hospitals performing pediatric surgery in participating Latin American countries.

We aim to assess the incidence of hospital postoperative complications in pediatric surgical patients < 18-years-old in Latin America. We will recruit all consecutive pediatric patients under the age of 18 years who were admitted to participating hospitals undergoing elective and nonelective surgery. The primary outcome is in-hospital postoperative complications up to 30 days after surgery.

DETAILED DESCRIPTION:
Background

Surgery is a cost-effective public health intervention. However, there are significant disparities in access to and in the safety of surgical and anesthesia services in low- and middle-income countries compared to high-income countries. (1) Additionally, there is a significant burden of surgical disease in the pediatric surgical population with a significant unmet need. (2,3) In Africa, children represent a significant proportion of the population, with approximately 50% of the population aged <19 years; moreover, this proportion is very similar in Latin America. (4) Postoperative complications are an important determinant of surgical morbidity and mortality. Limited data from Africa and Latin America suggest that risk factors, incidence, and outcomes associated with pediatric surgical complications differ in high-income countries. In the South African Pediatric Surgical Outcomes Study (SAPSOS), patients in this middle-income country (5) had twice the incidence of complications (6-8), and the types of complications differed from those in high-income countries, with a predominance of infectious complications. Furthermore, risk factors for complications (including ASA physical status, urgent surgery, surgery severity, and infectious indication for surgery) were different from those in high-income countries, wherein the risk factors include post-conceptual age, ASA physical status > 3, history of cardiovascular disease, and cardiovascular, neurological, or orthopedic surgical procedures. (9) Postoperative mortality was observed to be ten times higher in

South Africa than in a prospective study in high-income countries. (10) Furthermore, a prospective study of pediatric perioperative mortality in 24 Kenyan hospitals demonstrated a 7-day postoperative mortality of 1.7% (11), which is 17 times higher than that reported in high-income countries.

The African Surgical Outcomes Study (ASOS) described surgical outcomes in African adult patients. (12) Specifically, patients had a lower risk profile and fewer complications than those in high-income countries. However, postoperative mortality was twice the global average. A similar study is being performed in Latin America (LASOS), which also includes adults.

It is necessary to determine the importance of complications in pediatric surgical patients in Latin America, as well as the risk factors and types of complications that are experienced by these patients, due to the fact that data on this population are scarce. Consequently, we will be able to target appropriate interventions and funding to improve surgical outcomes for children in Latin America.

Study objectives

Primary objective

To determine the incidence of in-hospital postoperative complications up to 30 days after surgery in Latin American pediatric surgical patients (under 18-years-old).

Secondary objectives

In pediatric surgical patients under 18 years of age in Latin America, we aim to:

1. determine the perioperative in-hospital mortality rate up to 30 days after surgery;
2. determine the incidence of severe intraoperative adverse events;
3. determine the association between preoperative, intraoperative, and infrastructural factors and postoperative complications and death.

Methods

Study design

14-day Latin American international multicenter prospective cohort study of pediatric patients (<18 years) undergoing surgery.

Inclusion criteria

All of the consecutive patients under 18-years-old who were admitted to participating hospitals during the study period and who underwent elective and nonelective surgeries will be included in the study. This analysis will include outpatient surgeries and surgical procedures outside of operating rooms requiring local or general anesthesia. Recruitment will occur for fourteen days, starting on the date chosen by each participating hospital within the study cohort period (to be determined).

Exclusion criteria

1. patients undergoing radiological or other procedures that do not require general anesthesia or in which general anesthesia is performed but no procedure is performed (e.g., general anesthesia during MRI);
2. patients undergoing obstetric surgery.

Hospitals

Our goal is to recruit as many Latin American hospitals as possible. Each hospital will receive an individual report that compares its dataset with that of the overall national cohort.

Ethics in research and informed consent

Research ethics and regulatory approvals will be sought before the initiation of the study in each location by using national research legislation/guidelines for that country.

National leaders will ensure that the necessary ethical and regulatory approvals are obtained for participating hospitals in their country. Hospitals can only record data if there is ethical approval or an equivalent waiver.

This study is a large-scale clinical audit; therefore, it does not pose a significant risk to the study population. In most, if not all, countries, there will be no requirement for individual patient consent, as all of the data will be anonymized and are expected to be recorded as part of routine clinical practice.

A precedent has already been set from an international perspective. In the original EuSOS study, consent was provided in 27 of the 28 participating European countries. (13) In the ASOS study (12) and the ASOS-2 trial, consent was provided in most hospitals. In African pediatric perioperative studies, written informed consent was provided by six of eight ethics committees in the SAPSOS (5) study. Additionally, in a study in Kenya, written informed consent was provided in all 24 participating hospitals. (11) The LASOS study also obtained a consent form waiver from the coordinating center (Hospital das Clínicas HCFMUSP).

Informational signage documents will be used at participating sites to ensure that all of the patients and parents/guardians know that the hospital is participating in the study. These handover documents will be placed in critical areas of the participating hospitals, with explanations of the dates and nature of the study.

Recruitment and screening

We expect that all consecutive pediatric patients under 18 years undergoing elective and nonelective surgeries will be included in the study. Each hospital must record and submit a triage record of all of the eligible patients. Publicity through the appropriate hospital notices and signage will inform patients, their parents/guardians, and the public that the hospital is participating in the study.

Data collection and grouping

Each hospital will individually collect and record data on an electronic or paper case recording form (CRF) for each recruited patient. Paper CRFs will be stored in a locked office at each hospital, as they will include patient-identifiable data to allow for the tracking of clinical outcomes.

Data will be pseudoanonymized by generating a unique numeric code and transcribed by local investigators into a secure, password-protected electronic CRF on the REDCap platform. Each patient will be solely identified on the electronic CRF by their numerical code; thus, the study coordinating team can only trace the data back to an individual patient with contact with the local team. A participant (patient) list will be used at each hospital to match the identification codes in the database to individual patients to record clinical results and to provide any missing data points. Access to the data entry system will be protected by the username and password provided during the registration process to individual local investigators. All of the electronic data transfers between participating hospitals and the coordinating center will be encrypted by using a secure protocol (HTTPS/SSL 3.0 or higher).

When individual hospitals are unable to access the registration form over the internet, pseudoanonymous coded data can also be faxed, registered mailed, emailed, or WhatsApp messaged to the coordinating center (if necessary).

Each hospital will maintain a secure trial file, including a protocol, local investigator delegation record, ethics approval documentation, participant list, and other documentation (such as trial definitions).

A printout of the final summary of the included patients with essential variables should be produced for each hospital, along with the submission of final data for double-checking for completeness and accuracy.

Sample size calculation

We plan to recruit as many hospitals from each participating country as possible and ask them to include all eligible patients in the study. We do not have a specific sample size, and statistical models will be adapted to the event rate provided by the recruited sample to avoid inappropriate use of any logistic regression models.

Statistical analysis

The data to be collected are all collected as part of routine clinical care. Categorical variables will be described as proportions and compared by using chi-square tests. Continuous variables will be described as the mean and standard deviation if normally distributed or as the median and interquartile range if not normally distributed. The univariate analysis will test factors associated with postoperative complications, intensive care admission, and in-hospital death.

Hierarchical multilevel logistic regression models will be constructed to identify factors that are independently associated with these outcomes and to adjust for differences in confounding factors. Factors will be entered into the models based on their univariate relationship with the outcome (p<0.05), biological plausibility, and low rate of missing data. Logistic regression results will be reported as adjusted odds ratios (ORs) with 95% confidence intervals. Moreover, models will be evaluated by using sensitivity analyses to explore possible interacting factors and to examine any effect on the results. A statistical analysis plan will be written before the analysis.

Primary outcome

Postoperative complications in the hospital up to 30 days after surgery.

Secondary outcomes

1. Mortality on the day of surgery;
2. Hospital mortality up to 30 days after surgery;
3. Risk factors associated with in-hospital complications;
4. Severe intraoperative critical adverse events;
5. Level of qualification of anesthesia and surgery providers, as well as the number of specialists per pediatric population;
6. Admission to intensive care.

ELIGIBILITY:
Inclusion Criteria:

* All of the consecutive patients under 18-years-old who were admitted to participating hospitals during the study period and who underwent elective and nonelective surgeries will be included in the study.

Exclusion Criteria:

1. patients undergoing radiological or other procedures that do not require general anesthesia or in which general anesthesia is performed but no procedure is performed (e.g., general anesthesia during MRI);
2. patients undergoing obstetric surgery.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children submitted to surgery (elective and non-elective).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative in-hospital complication | until 30 days
  Percentage of postoperative complications in-hospital

SECONDARY OUTCOMES:
Surgical mortality | until 30 days
  Percentage of surgical mortality in-hospital
Admission to critical care | until 30 days
  Percentage of children admitted in critical care

CONTACTS AND LOCATIONS:
Overall Officials: Vinicius Quintao, MD, PhD, Principal Investigator — Postdoctoral fellow
Locations (1):
- Academic Reserach Organization, Instituto do Coracao, Hospital das Clinicas, Faculdade de Medicina, Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bainbridge D, Martin J, Arango M, Cheng D; Evidence-based Peri-operative Clinical Outcomes Research (EPiCOR) Group. Perioperative and anaesthetic-related mortality in developed and developing countries: a systematic review and meta-analysis. Lancet. 2012 Sep 22;380(9847):1075-81. doi: 10.1016/S0140-6736(12)60990-8. PMID 22998717
- [Result] Bickler SW, Rode H. Surgical services for children in developing countries. Bull World Health Organ. 2002;80(10):829-35. Epub 2002 Nov 28. PMID 12471405
- [Result] Butler EK, Tran TM, Nagarajan N, Canner J, Fuller AT, Kushner A, Haglund MM, Smith ER; SOSAS 4 Country Research Group. Epidemiology of pediatric surgical needs in low-income countries. PLoS One. 2017 Mar 3;12(3):e0170968. doi: 10.1371/journal.pone.0170968. eCollection 2017. PMID 28257418
- [Result] Torborg A, Cronje L, Thomas J, Meyer H, Bhettay A, Diedericks J, Cilliers C, Kluyts H, Mrara B, Kalipa M, Rodseth R, Biccard B; South African Paediatric Surgical Outcomes Study Investigators. South African Paediatric Surgical Outcomes Study: a 14-day prospective, observational cohort study of paediatric surgical patients. Br J Anaesth. 2019 Feb;122(2):224-232. doi: 10.1016/j.bja.2018.11.015. Epub 2018 Dec 19. PMID 30686308
- [Result] GlobalSurg Collaborative. Determinants of morbidity and mortality following emergency abdominal surgery in children in low-income and middle-income countries. BMJ Glob Health. 2016 Dec 12;1(4):e000091. doi: 10.1136/bmjgh-2016-000091. eCollection 2016. PMID 28588977
- [Result] Habre W, Disma N, Virag K, Becke K, Hansen TG, Johr M, Leva B, Morton NS, Vermeulen PM, Zielinska M, Boda K, Veyckemans F; APRICOT Group of the European Society of Anaesthesiology Clinical Trial Network. Incidence of severe critical events in paediatric anaesthesia (APRICOT): a prospective multicentre observational study in 261 hospitals in Europe. Lancet Respir Med. 2017 May;5(5):412-425. doi: 10.1016/S2213-2600(17)30116-9. Epub 2017 Mar 28. PMID 28363725
- [Derived] Quintao VC, de Sousa GS, Torborg A, Vieira A, Consonni F, Rodrigues S, Proenca J, Carlos RV, Clemente M, Alonso N, Neville M, Leite F, Tonello C, Evans F, Garcia-Marcinkiewicz A, Guris R, Herrera J, Andersen A, Schaigorodsky L, Biondini N, Cajas N, Cruzat F, Cortinez LI, Giraldo M, Valle A, Pozo C, Betancourt A, Echeto MA, Dominguez A, Sarmiento L, Gonzalez K, Abrego G, Leguizamon L, Paula L, Lauber C, Lopez G, Biccard BM, Carmona MJ, Hajjar LA. Latin American Surgical Outcomes Study in Paediatrics (LASOS-Peds): study protocol and statistical analysis plan for a multicentre international observational cohort study. BMJ Open. 2024 Sep 23;14(9):e086350. doi: 10.1136/bmjopen-2024-086350. PMID 39313281